CLINICAL TRIAL: NCT06126588
Title: Combination of Everolimus and 177Lu-DOTATATE in the Treatment of Grades 2 and 3 Refractory Meningioma: a Phase IIb Clinical Trial
Acronym: ELUMEN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Principal Investigator, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021PI203
Record Dates: First submitted 2023-10-27; First posted 2023-11-13 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient treat with everolimus (Experimental): The product Everolimus is an oral drug.The dosage is 7.5 mg.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Patient will be treat during 7 months of Everolimus

SUMMARY:
Meningioma, the most common intracranial primary tumor of the central nervous system predominantly affects people in their fifties. Meningiomas are generally subdivided into two entities: a priori non-aggressive meningiomas (grade 1), and meningiomas at high risk of aggressive behavior (grade 2/atypical and 3/anaplastic). The current conventional treatments for meningioma are surgery and radiotherapy. When these treatments are no longer feasible, meningiomas are considered refractory irrespectively of grade, and in these rare entities, the therapeutic arsenal is reduced to the few treatments that have shown limited efficacy. Refractory, and particularly grades 2 and 3 meningiomas, have very poor prognoses with a progression-free survival at 6 months (PFS-6) of 26%. The European Response Assessment in Neuro-Oncology group (RANO) recommends that in any new, grades 2 and 3 meningioma, therapy that achieves a PFS-6 >30% in phase II trials be considered promising.

In Nuclear Medicine, Peptide Receptor Radionuclide Therapy (PRRT) with 177Lu-DOTATATE, currently used on a compassionate basis in refractory meningioma, deploys an octreotide-like effect, and appears very promising, with preliminary PFS-6 of 94% and an overall survival at 12 months (OS-12) of 88% in grade 1 meningioma. However, its PFS-6 is reduced to 28% with an OS-12 of 65% in WHO grades 2 and 3 meningioma. Recently the non-radiolabeled octreotide and everolimus combination however achieved a PFS-6 of 55% and an OS-12 of 75% in a population of 90% WHO grades 2 and 3 meningioma.

DETAILED DESCRIPTION:
Meningioma, the most common intracranial primary tumor of the central nervous system predominantly affects people in their fifties. Meningiomas are generally subdivided into two entities: a priori non-aggressive meningiomas (grade 1), and meningiomas at high risk of aggressive behavior (grade 2/atypical and 3/anaplastic). The current conventional treatments for meningioma are surgery and radiotherapy. When these treatments are no longer feasible, meningiomas are considered refractory irrespectively of grade, and in these rare entities, the therapeutic arsenal is reduced to the few treatments that have shown limited efficacy. Refractory, and particularly grades 2 and 3 meningiomas, have very poor prognoses with a progression-free survival at 6 months (PFS-6) of 26%. The European Response Assessment in Neuro-Oncology group (RANO) recommends that in any new, grades 2 and 3 meningioma, therapy that achieves a PFS-6 >30% in phase II trials be considered promising.

In Nuclear Medicine, Peptide Receptor Radionuclide Therapy (PRRT) with 177Lu-DOTATATE, currently used on a compassionate basis in refractory meningioma, deploys an octreotide-like effect, and appears very promising, with preliminary PFS-6 of 94% and an overall survival at 12 months (OS-12) of 88% in grade 1 meningioma. However, its PFS-6 is reduced to 28% with an OS-12 of 65% in WHO grades 2 and 3 meningioma. Recently the non-radiolabeled octreotide and everolimus combination however achieved a PFS-6 of 55% and an OS-12 of 75% in a population of 90% WHO grades 2 and 3 meningioma.

Our research hypothesis is that 177Lu-DOTATATE PRRT, a vector targeting somatostatin type 2 receptor (octreotide type) with a high-energy β-emitting radioactive label, when combined with everolimus, an mTOR protein inhibitor with radiosensitizing properties, will potentiate the effects of the non-radiolabeled octreotide + everolimus combination and increase PFS-6 in refractory grades 2 and 3 meningioma patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient < 80 years old, who received a complete comprehensive briefing about the trial and signed the informed consent
* Eligible patient for compassional access program (National Multidisciplinary Neuro-Oncology board to Lutathera ® traitement
* WHO performance status ≤ 3
* Patient with grade 2 and 3 meningioma, substantiated by histology, not amenable to surgery or radiotherapy, with clinical or radiological progression
* Clinical deterioration or at least 10% of tumor growth rate, defined as the product of the two largest diameters of the target lesion within 6 months
* Expressing somatostatin receptors as determined by 68Ga-DOTATOC PET (lesion uptake ≥ liver uptake and/or 1.7 fold SUVpeak of the controlateral meninges).
* Patient that underwent a brain MRI and 68Ga-DOTATOC PET within the last 2 months.
* Effective contraception required for women of childbearing age.
* Patient with social security cover.

Exclusion Criteria:

* Hypersensitivity to everolimus.
* Contraindication to 177Lu-DOTATATE: renal failure GFR<40 mL/min/1.73m2 (calculated by the CKD-Epi Formula), hepatic failure total bilirubin >3N, heart failure NYHA III or IV.

Patients should not take the following treatments:

* Other rapamycin derivatives (sirolimus, temsirolimus, deforolimus).
* Other immunosuppressants
* Co-administration with potent inhibitors and inducers of CYP3A4 and/or the multidrug efflux pump P-glycoprotein (PgP) : Ketoconazole , itraconazole, posaconazole, voriconazole, telithromycin, clarithromycin, Nefazodone, Ritonavir, atazanavir, saquinavir, darunavir, indinavir, nelfinavir.
* If everolimus is taken with orally administered CYP3A4 substrates with a narrow therapeutic index (e.g. pimozide, terfenadine, astemizole, cisapride, quinidine or ergot alkaloid derivatives), the patient should be monitored for undesirable effects described in the product information of the orally administered CYP3A4 substrate.
* Contraindication to MRI or 68Ga-DOTATOC PET/CT.
* Person referred to and L. 3212-1 and L. 3213-1 (psychiatric care).
* Women of childbearing age without effective contraception
* Patient unable to attend follow-ups over a 12-month period.
* Patients who participate in an interventional clinical research trial for the duration of the ELUMEN study.
* Individuals referred to in Articles 10, 31, 32, 33 and 34 of Regulation (EU) No 536/2014.
* Pregnant woman, birthing or breastfeeding mother
* Minor (not emancipated)
* Adult subject to a legal protection measure (such as guardianship, conservatorship)
* Adult who is unable to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
RANO criteria (Response assessment in neuro oncology criteria) | 7 months
  Progression Free Survival (PFS) from the start of treatment according to the RANO criteria (Response assessment in neuro oncology criteria)

SECONDARY OUTCOMES:
Overall Survival | 12 months
  OS-12. Overall Survival, defined as the time from the date of inclusion to the date of death from any cause
Tumor growth rate | 6 months
  Tumor growth rate, defined as the product of the two largest diameters of the target lesion from the MRI (Magnetic Resonance Imaging) at Month 3 or Month 6 compared to the diameters of the lesion at baseline.
Progression Free Survival | 1 month
  Dose delivered to the tumor (dosimetry) will be calculated on at least 2 skull scans with 177Lu-DOTATATE SPECT-CT (D1 and D7), after the first cycle of 177Lu-DOTATATE.
Number and types of grade 1, 2, 3 or 4 adverse events according to the CTCAE | 180 days
  Number and types of grade 1, 2, 3 or 4 adverse events according to the CTCAE (Common Terminology Criteria for Adverse Events) classification per patient, from the start of treatment until 180 days after the end of the last treatment cycle.
Questionnaire | 6 moniths
  HRQoL (Measuring Health-related quality of life ), assessed using the EORTC (uropean Organisation for Research and Treatment of Cancer) QLQ-C30 (Quality of Life Control) questionnaire at inclusion (V1) and at 6 months (V7).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU of Nancy, Vandœuvre-lès-Nancy, Grand Est
  - Nancy Hospital, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No